CLINICAL TRIAL: NCT06114355
Title: Comparison of Pre-operative EUS Guided and Intra-operative Direct Portal Vein Pressure Measurement in Pretransplant Cirrhotics - Prospective Observational Study
Brief Title: Comparison of Pre-operative EUS Guided and Intra-operative Direct Portal Vein Pressure Measurement in Pretransplant Cirrhotics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant, Asian Institute of Gastroenterology, India
Other Study IDs: PV01
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: EUS Portal pressure measurement — Direct portal pressure measurement under EUS-guidance (EUS-PPM) is a promising alternative to conventional indirect Hepatic Venous Pressure Gradient (HVPG). In patients undergoing liver transplantation for cirrhosis, high pre-operative portal vein (PV) pressure requires intra-operative portal vein inflow modulation (PIM)

SUMMARY:
Direct portal pressure measurement under EUS-guidance (EUS-PPM) is a promising alternative to conventional indirect Hepatic Venous Pressure Gradient (HVPG). In patients undergoing liver transplantation for cirrhosis, high pre-operative portal vein (PV) pressure requires intra-operative portal vein inflow modulation (PIM). This pilot study aims to assess correlation between EUS-PPM with direct intra-operative portal pressure measurement (IO-PPM).

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis patients scheduled for liver transplant for the standard indications within next 24- 48 hours will be included.

Exclusion Criteria:

* Severe ascites not amenable for tapping
* History of blood thinner consumption within last 5 days
* Active duodenal ulcerations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decompensated Cirrhosis patient listed for liver transplant according to the standard indications.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between EUS-PPM with direct intra-operative portal pressure measurement (IO-PPM). | 1 year
  Correlation between EUS-PPM with direct intra-operative portal pressure measurement (IO-PPM).

SECONDARY OUTCOMES:
Correlation between readings of EUS-PPM using portable manometry set and arterial transducer. | 1 year
  Correlation between readings of EUS-PPM using portable manometry set and arterial transducer.